CLINICAL TRIAL: NCT05384574
Title: Vitamin D Supplementation and Clinical Outcomes in Severe COVID-19 Patients - Randomized Controlled Trial
Brief Title: Vitamin D Supplementation and Clinical Outcomes in Severe COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Lenko Saric, Anesthesiology and Intensive Care specialist, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2181-147/01/06/M.S.-21-02
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Covid-19; Respiratory Distress Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients with low levels of Vitamin D on admission to ICU randomized to receive vitamin D supplementation
  Interventions: Dietary Supplement: cholecalciferol
- Control (No Intervention): Patients with low levels of Vitamin D on admission to ICU not receiving vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: cholecalciferol — daily supplementation of cholecalciferol, 10 000 IU, during 14 days
  Arms: Intervention

SUMMARY:
Single center, open label randomized clinical trial.

Study location: tertiary hospital center (University Hospital Split, Croatia). All COVID-19 patients with positive PCR test admitted to ICU and in need for respiratory support will be eligible for inclusion in this study.

Patients admitted to ICU with severe COVID-19 disease and in need for invasive or non-invasive respiratory support with low levels of vitamin D (<50 nmol/l) measured on admission. All patients are older than 18 years and have confirmed COVID-19 disease with PCR test.

Intervention:

All patients included in this study will receive standard of care. Patients randomized into intervention group will be receiving 10 000 IU of cholecalciferol daily. Supplement will be administered orally or via gastric tube during ICU stay or for at least 14 days in case of ICU discharge before day 14. Supplementation will begin within 48 hours of admission to ICU. Supplement will be prepared and administered by experienced nursing staff. For patients receiving supplementation, vitamin D levels will be checked on days 7 and 14. In case that vitamin D levels are > 150 nmol/l or if the calcium levels are consistently > 2.6 mmol/l, further supplementation will be stopped.

Outcomes:

Primary outcome is number of days spent on ventilator.

Secondary outcomes: all-cause mortality on day 28, all-cause mortality on day 60, mortality at hospital discharge, clinical improvement at day 28 (WHO clinical progression scale), days spent in ICU, days spent in hospital after discharge from ICU, need for dialysis at day 28, bacterial superinfections, neutrophile to lymphocyte ratio, disease severity (CRP levels, PaO2/FiO2 ratio, D-dimer levels, fibrinogen, ferritin, PCT), adverse outcomes.

Hypothesis: patients receiving Vitamin D supplementation will have shorter number of days spent on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU with severe COVID-19 disease and in need for invasive or non-invasive respiratory support with low levels of vitamin D (<50 nmol/l) measured on admission. All patients are older than 18 years and have confirmed COVID-19 disease with PCR test.

Exclusion Criteria:

* Patients will be excluded from study in case of calcium levels that are consistently above normal serum range (> 2.6 mmol/L, > 10.5 mg/dL) or if vitamin D levels are > 150 nmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
number of days on mechanical ventilation | Daily, through study completion, on average 6 months
  Number of days spent on mechanical ventilation for each patient

SECONDARY OUTCOMES:
All-cause mortality on day 28 | day 28
  Number of patients alive on day 28
All-cause mortality on day 60 | day 60
  Number of patients alive on day 60
clinical improvement at day 28 | day 28
  World Health Organization Clinical progression scale. Values are from 0 to 10 with higher score meaning worse clinical status
Number of days spent in ICU | Daily, through study completion, on average 6 months
  Number of days spent in Intensive care unit for each patient
Number of days spent in hospital after ICU discharge | Daily, through study completion, on average 6 months
  Number of days spent in hospital for each patient
Acute renal failure | Day 28
  Number of patients with need for renal replacement therapy
bacterial superinfections | Daily, through study completion, on average 6 months
  Number of patients with bacterial superinfections during hospitalization
CRP levels (mg/ml) | Daily, through study completion, on average 6 months
  blood tests will be taken daily during hospital stay
prokalcitonin levels (ng/ml) | Daily, through study completion, on average 6 months
  blood tests will be taken daily during hospital stay
fibrinogen levels (g/L) | Daily, through study completion, on average 6 months
  blood tests will be taken daily during hospital stay
D-dimer levels (mg/l) | Daily, through study completion, on average 6 months
  blood tests will be taken daily during hospital stay
adverse outcomes | Daily, through study completion, on average 6 months
  Number of patients with elevated serum calcium levels

CONTACTS AND LOCATIONS:
Overall Officials: Lenko Saric, M.D. PhD, Principal Investigator — University Hospital Split, Croatia
Locations (1):
- University Hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No